CLINICAL TRIAL: NCT02735720
Title: The CardiOvascular Remodeling Following Endovascular Aortic Repair (CORE) Study
Acronym: CORE
Status: Terminated | Type: Observational
Why Stopped: Because of the difficulties created by COVID-19 and bringing participants on onsite, the decision was made to stop recruitment.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alberto Figueroa, Principal Investigator, University of Michigan
Other Study IDs: CORE01
Record Dates: First submitted 2016-03-28; First posted 2016-04-13 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: thoracic endovascular aortic repair; endograft; cardiac remodelling; thoracic aortic aneurysm; penetrating aortic ulcer; MRI
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood testing will include complete blood count with platelets (including white blood cells, hemoglobine, hematocrit, red blood cells), a basic metabolic panel (including sodium, potassium, glucose, and calcium. Cardiac biomarkers testing will include natriuretic peptide (BNP), amino-terminal pro-BNP (NT-pro-BNP) and Troponin T.
  The investigators will not determine DNA of the patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TEVAR group: Adult patients whose clinician's are managing their thoracic aortic aneurysms or with penetrating aortic ulcers with TEVAR.
  Standard work-up examinations for TEVAR will be collected, consisting of computed tomography (CT), echocardiography, blood pressure, heart rate, ECG and blood tests. Prior to the TEVAR procedure, a non-invasive MRI scan and blood samples will be acquired. Intraoperative pressure measurements will be collected during the TEVAR. One year following TEVAR, the subject will undergo a second non-invasive MRI study in addition to the standard clinical imaging follow-up CT-scan. Measurements of blood pressure, heart rate, ECG, and blood testing will also be repeated at follow-up.
  Interventions: Other: TEVAR; Other: Non-TEVAR medical treatment
- Non-TEVAR medical treatment group: Adult patients whose clinician's are managing their thoracic aortic aneurysms or with penetrating aortic ulcers with pharmacological treatment alone.
  Patients with stable thoracic aortic aneurysms or with penetrating aortic ulcers not requiring aortic repair are monitored in the outpatient clinic as standard of care. The investigators will collect blood pressures and heart rates in these patients, which are acquired as standard of care. In addition, in this study, these subjects will undergo an ECG, blood testing and one non-invasive MRI scan at baseline. One year after baseline, this group will undergo a second non-invasive MRI study, with subsequent blood pressure and heart rate measurements, ECG and blood testing.
  Interventions: Other: Non-TEVAR medical treatment

INTERVENTIONS:
Other: TEVAR — Thoracic endovascular aortic repair, which includes the implantation of stent-graft in the thoracic aorta to repair the lesion. This may be done with a variety of stent-graft brands and types. The type and brand of stent-graft is left to the discretion of the care taking physician.
  Groups: TEVAR group
Other: Non-TEVAR medical treatment — Any clinical management by physicians caring for these patients. This includes whatever blood pressure and heart rate medication is prescribed by the treating physician, without any surgery. The type and dosage of medication is left to the discretion of the care taking physician.

SUMMARY:
The use of TEVAR is increasing rapidly and patients even in younger patients. However, current endografts are several orders of magnitude stiffer than the native aorta. Pre-clinical and clinical studies have reported acute aortic stiffening after TEVAR resulting in hypertension, elevated pulse pressure, cardiac remodeling, reduced coronary perfusion, and finally, heart failure. These effects are markedly profound in young patients, as their hearts and aortas are more compliant. Previous studies on adverse cardiovascular remodeling have important limitations, such as retrospective design, use of echocardiography (with low reproducibility and high operator-dependency), and mixed populations. A systematic assessment of the deleterious effects of TEVAR is still missing.

The objective of this study is to perform a prospective, non-randomized controlled, study in which blood pressure, heart rate, ECG, echocardiography, CT, MRI, intra-luminal hemodynamic assessment, computational modeling and biomarkers are used to assess cardiovascular remodeling following TEVAR. This study targets patients with thoracic aortic aneurysms (TAA) or penetrating aortic ulcers (PAU) treated with TEVAR. A control group will consist of TAA and PAU subjects who do not require endovascular treatment.

The specific aims of the study include: 1) Quantification of cardiovascular remodeling following TEVAR in TAA or PAU patients. 2) Validation of computational modeling of thoracic aortic hemodynamics following TEVAR using the above clinical measurements. Once validated, computational analyses will be performed to virtually assess the impact of more compliant endografts on cardiac and aortic hemodynamics. 3) Investigation of diagnostic accuracy of ECG, BNP, NT-pro-BNP and Troponin T, for cardiac remodeling compared to MRI, the reference method.

This study will assess the impact of thoracic aortic stent grafts on the cardiovascular system through non-invasive measurements. Although there are no direct benefits for the enrolled subjects, future aortic patients might benefit from better patient management with improved aortic endograft designs and long-term outcomes.

DETAILED DESCRIPTION:
Patient Population and Clinical Measurements:

The Frankel Cardiovascular Center at the University of Michigan Health System (UMHS) is a regional center with expertise in managing a large variety of aortic diseases. Only adult patients (age between 18-99 years) will be included. Patients will be included regardless of race or ethnicity. The patient population consists of:

1. Patients with a descending thoracic aortic aneurysm (TAA). TAA is defined by a balloon-like dilatation of the thoracic aorta. Such a dilatation may grow and eventually rupture, associated with high mortality. In the United States, more than 10,000 patients die every year due to a ruptured aneurysm. Current United States guidelines state that when the diameter of a TAA in patients with no connective tissue disorder is larger than 55-60 mm, aortic repair is recommended. To date, TEVAR is the first choice of therapy unless the anatomy is unsuitable or the patient has a connective tissue disorder.
2. Patients with a penetrating aortic ulcer (PAU). PAU is a chronic aortic condition, defined by an ulcer-like disruption of the inner aortic wall. Up to 28% of patients with a PAU may have or may develop an aortic aneurysm. Treatment with TEVAR is recommended for these patients, especially when patients are complicated by aortic growth or rupture.

Study Design:

TEVAR Group. In this study, the investigators target both TAA and PAU treated with TEVAR. Patients are to be identified in the clinic setting. Patients who are planned for treatment TEVAR for TAA and PAU (based on their treating physician's decision) will be given information about this observational study. Results for the standard work-up examinations for TEVAR, which consist of computed tomography (CT), echocardiography, blood (BP) and heart (HR) measurements, and electrocardiogram (ECG) will be collected. Once patient consent is confirmed, and prior to the TEVAR procedure, this study will include a non-invasive MRI scan and a blood collection for the biomarker data, in addition to the standard of care. In this study, during the TEVAR procedure, intraluminal pressure measurements will be conducted using the catheters and guidewires that will be already in place for the deployment of the endograft. This study will neither delay or modify their endovascular procedure. One year (between a window of 275 - 455 days) following the TEVAR procedure, the subject will undergo and a second non-invasive MRI study in addition to the standard clinical imaging follow-up. During this follow-up imaging, the patients will also undergo BP and HR measurements, ECG and blood tests.

Control Group. Patients with a stable TAA or PAU who do not require surgery are monitored in the outpatient clinic as standard of care. In this study, these patients will be given information about our study and will be asked to be included in our investigation. Once consent of the patients is confirmed, participants will undergo BP and HR measurements, ECG, blood tests, and one non-invasive MRI scan, at baseline. One year (between a window of 275 - 455 days) after baseline, the participants will undergo additional observations; non-invasive MRI study, BP and HR measurements, ECG and blood tests.

Clinical Measurements:

BP, HR, ECG, and blood- tests will be collected by trained personnel on all at baseline, and at one year (between a window of 275 - 455 days) follow-up.

* BP and HR will be measured per standard protocol.
* ECG will consist of a standard 12 lead ECG.
* Standard blood tests include complete blood count with platelets (including white blood cells, hemoglobin, hematocrit, red blood cells), a basic metabolic panel (including sodium, potassium, glucose, and calcium. Cardiac biomarkers tests include natriuretic peptide (BNP), amino-terminal pro-BNP (NT-pro-BNP) and Troponin T.

Echocardiography - Preoperative echocardiography is standard of care in all patients requiring TEVAR. The obtained echocardiographic measurements in these patients will be collected and compared to the preoperative MRI data.

Intraluminal pressures - During TEVAR, an angiography will be performed as standard of care. In this study, intraluminal pressure measurements will be conducted in the TEVAR group, using the catheters and guidewires that will be already in place for the deployment of the endograft, as is commonly done at the UMHS.

MRI - This study will employ the following clinical and (FDA/IRB approved) research MRI sequences to assess multiple signs of cardiovascular remodeling:

Clinical sequences:

1. Phase-contrast MRI measurements will be acquired on different cross-sections of the aorta (through-plane velocity-encoding). Images will also be captured in an oblique sagittal view (in-plane velocity-encoding) to estimate the aortic vessel wall stiffness via pulse wave velocity measurements. Velocity-encoded phase-contrast MRI images will be acquired across the mitral valve to evaluate the left ventricular (LV) diastolic function through the measurement of early-to-atrial ratios. Myocardial perfusion images will be acquired after administration of gadolinium based contrast agent under pharmacological stress.
2. Cine measurements will include LV volume, LV wall volume and left atrial volume.
3. Tag-MRI will measure different components of myocardial strain in standard short-axis and four-chamber views.

Research sequences:

1. Strain encoding sequences will measure cardiac- and aortic strain. This sequence is IRB approved: IRBMED # 2004-0452.
2. Steady state free precession sequences will measure strain of the thoracic aorta through cine measurements in the ascending aorta just distal to the coronary branches and just proximal to the celiac trunk. The sequence is obtained in accordance within FDA safety guidelines and with FDA approved MRI machines. It is easily reproducible and quantifiable and confirms to all MRI safety parameters in the United States.

All these measurements are non-invasive and therefore do not impose additional risk or burden to the patient. Contrast will be administered, except for those patients with poor renal function (eGFR<60). The total anticipated scan time is approximately 1 hour.

Computational Modeling - Using the imaging and clinical data, simulations of blood flow and pressure will be performed using computational fluid dynamics (CFD) techniques and the High-Performance Computer cluster "Flux" at the University of Michigan. Highly detailed descriptions of velocity, flow, pressure, wall shear stress and other hemodynamically significant quantities will be obtained. The results of these non-invasive simulations will be compared against the clinical measurements (BP, HR, echocardiography, MRI, and intraluminal pressures) to calibrate this tool. Once calibrated, computational analyses will be performed to virtually assess the impact of more compliant endografts on cardiac and aortic hemodynamics.

Statistical Analysis - Statistical analysis will include descriptive and comparative analysis of both clinical measurements and data acquired from computational modeling. In analysis, participants will be grouped by TEVAR or Control group. Sub-analysis will include grouping by endograft length, gender, and age. The patients identifying information and protected health data will be dealt with based on HIPAA guidelines.

Preliminary echocardiographic data of TAA patients treated with TEVAR at the University of Michigan Health System revealed an average LV mass increase of 39% (P = 0.047) at 1-year follow-up. Power analysis for a Mann-Whitney U test, based on these preliminary data, calculated that for a significant threshold of 5% (P < 0.05, two-sided test) a total sample size of 20 patients (α = 0.05, power = 97%) would be needed to observe a significant effect of TEVAR on LV mass increase. To ensure a margin of error, the investigators aim to include 12 TEVAR patients and 12 control patients.

To sum up, the end-goal of this study is to assess the impact of TEVAR on adverse cardiovascular remodeling through imaging and computation. This impact remains unclear and may carry important implications for patient management and future endograft design. The additional measurements required for this study are almost risk-free for all included participants. Although there are no direct benefits for the enrolled subjects, future aortic patients might benefit from better patient management with improved aortic endograft designs and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with descending thoracic aortic aneurysms or with penetrating aortic ulcers.
* Subject willing to return for one year follow up and comply with protocol requirements.

Exclusion Criteria:

* Ejection fraction < 35%; LV wall motion abnormality
* Poor renal function (estimated glomerular filtration rate (eGFR) < 60 mL/min/173 m2)
* Pregnancy
* Connective tissue disorder
* Significant valve, lung or congenital heart disease
* History of cardiac or aortic surgery
* Expected cardiac or aortic surgery within the study period
* Standard MRI contraindications (pacemakers, non-compatible metal implants, and claustrophobia)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will consist of adult patients with descending thoracic aortic aneurysms or with penetrating aortic ulcers managed with TEVAR (TEVAR group, n=12) or with optimal medical treatment alone (control group, n=12) at the University of Michigan Health System.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular mass (g), quantified with cardiac MRI | 1 year
  This will be quantified in grams.

SECONDARY OUTCOMES:
Diagnostic accuracy of ECG for cardiac remodelling compared to MRI | 1 year
  A standard 12-lead ECG will be obtained and left ventricular hypertrophy will be assessed (i.e. QRS complex widening, abnormal ST segments or T waves).
Diagnostic accuracy of ECG alone, and in combination with BNP, NT-pro-BNP, and Troponin T for cardiac remodelling compared to MRI | 1 year
  A standard 12-lead ECG will be obtained and left ventricular hypertrophy will be assessed (i.e. QRS complex widening, abnormal ST segments or T waves).
  Cardiac biomarkers BNP, NT-pro-BNP, and Troponin T will be quantified in blood samples.
Validation of computational modelling of thoracic aortic hemodynamics (i.e. velocity, flow, and pressure) following TEVAR against intra-luminal pressures and MRI. | 1 year
  Hemodynamics (i.e. velocity in ml/min, flow in mm3/min, and pressure in mmHg) measured with intraluminal catheters and MRI will be used to create and validate patient-specific computational models. Subsequently, the impact of more compliant stent-grafts on aortic hemodynamics will be assessed.
Early-to-late atrial filling ratios measured through cardiac MRI | 1 year
  Early-to-late atrial filling ratios of the left atrium will be quantified using cardiac MRI.
Aortic flow (ml/min) measured through cardiac MRI | 1 year
  Aortic flow (ml/min) will be quantified using phase-contrast MRI at the intersections of the ascending aorta, all arch branches, proximal descending aorta, and distal descending aorta.
Myocardial strain (%) using MRI sequences. | 1 year
  Strain-encoding (SENC) or conventional tagged images will be used to quantify cardiac strain (%) at the basal, mid-ventricular, and apical short-axis slices, as well as in a 4-chamber slice.
Central aortic pulse wave velocity using phase-contrast MRI. | 1 year
  Phase-contrast MRI measurements will be acquired at different levels of the thoracic aorta using through-plane velocity-encoding and in an oblique sagittal view (in-plane velocity-encoding) to estimate the aortic vessel wall stiffness via PWV (cm/s) measurements.
Myocardial perfusion using MRI perfusion sequences. | 1 year
  Myocardial perfusion images will be acquired after administration of gadolinium-based contrast agent under pharmacological stress. The investigators will determine perfusion defects as well as the myocardium contrast uptake (ml/min/g) and contrast washout curves.
Aortic strain (%) using MRI sequences. | 1 year
  Cine images will be used to measure strain (%) of the thoracic aorta through measurements in the ascending aorta just distal to the coronary branches and proximal to the celiac trunk.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto C Figueroa, PhD, Principal Investigator — Departments of Biomedical Engineering and Surgery, University of Michigan, USA
Locations (1):
- Department of Cardiac Surgery, University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takeda Y, Sakata Y, Ohtani T, Tamaki S, Omori Y, Tsukamoto Y, Aizawa Y, Shimamura K, Shirakawa Y, Kuratani T, Sawa Y, Yamamoto K, Mano T, Komuro I. Endovascular aortic repair increases vascular stiffness and alters cardiac structure and function. Circ J. 2014;78(2):322-8. doi: 10.1253/circj.cj-13-0877. Epub 2013 Nov 29. PMID 24292128
- [Background] Tzilalis VD, Kamvysis D, Panagou P, Kaskarelis I, Lazarides MK, Perdikides T, Prassopoulos P, Boudoulas H. Increased pulse wave velocity and arterial hypertension in young patients with thoracic aortic endografts. Ann Vasc Surg. 2012 May;26(4):462-7. doi: 10.1016/j.avsg.2011.06.021. Epub 2012 Jan 27. PMID 22284778
- [Background] Roccabianca S, Figueroa CA, Tellides G, Humphrey JD. Quantification of regional differences in aortic stiffness in the aging human. J Mech Behav Biomed Mater. 2014 Jan;29:618-34. doi: 10.1016/j.jmbbm.2013.01.026. Epub 2013 Feb 9. PMID 23499251
- [Background] Coogan JS, Humphrey JD, Figueroa CA. Computational simulations of hemodynamic changes within thoracic, coronary, and cerebral arteries following early wall remodeling in response to distal aortic coarctation. Biomech Model Mechanobiol. 2013 Jan;12(1):79-93. doi: 10.1007/s10237-012-0383-x. Epub 2012 Mar 14. PMID 22415052
- [Result] Nauta FJ, Kamman AV, Ibrahim EH, Agarwal PP, Yang B, Kim K, Williams DM, van Herwaarden JA, Moll FL, Eagle KA, Trimarchi S, Patel HJ, Figueroa CA. Assessment of CardiOvascular Remodelling following Endovascular aortic repair through imaging and computation: the CORE prospective observational cohort study protocol. BMJ Open. 2016 Nov 17;6(11):e012270. doi: 10.1136/bmjopen-2016-012270. PMID 27856475
- [Result] van Bakel TMJ, Arthurs CJ, Nauta FJH, Eagle KA, van Herwaarden JA, Moll FL, Trimarchi S, Patel HJ, Figueroa CA. Cardiac remodelling following thoracic endovascular aortic repair for descending aortic aneurysms. Eur J Cardiothorac Surg. 2019 Jun 1;55(6):1061-1070. doi: 10.1093/ejcts/ezy399. PMID 30535179
- [Result] van Bakel TMJ, Burris NS, Patel HJ, Figueroa CA. Ascending aortic rupture after zone 2 endovascular repair: a multiparametric computational analysis. Eur J Cardiothorac Surg. 2019 Sep 1;56(3):618-621. doi: 10.1093/ejcts/ezy458. PMID 30608518
- See also: Computational lab where computational modeling will be conducted — http://bloodflow.engin.umich.edu/